CLINICAL TRIAL: NCT05017636
Title: Mechanical and Physiological Effect of Noncorporeal Shock Wave Therapy Without Biological Stress-histological and Immuno-histochemical Analysis
Brief Title: Effect of Shock Wave Therapy Without Biological and Immuno-histochemical Analysis.
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: shock wave
Record Dates: First submitted 2019-10-29; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: fat localized; sagging skin; Obesity
MeSH Terms: conditions — Obesity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: experimental study
Masking Description: N/D
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment groupThorck Shock Wave Ibramed (terapia ESWT)- fat cell death (Active Comparator): The shock wave treatment was performed on the left side of the abdomen
  Interventions: Device: shock wave therapy
- Without intervention. (No Intervention): no shockwave treatment was performed on the right side of the abdomen, which was specified as a control group no shockwave treatment was performed on the right side of the abdomen, which was specified as a control group without intervention.

INTERVENTIONS:
Device: shock wave therapy — The participants received the treatment protocol established by the manufacturer of the Thork Shock Wave® device, IBRAMED- Industria Brasileira de Equipamentos Electromédicos, Amparo, São Paulo approved by Anvisa No. 10360310036. (Figure 1). The parameters were, 4,000 thousand shots with energy of 180mJ and frequency of 15Hz with 15mm stainless steel tip and 2,000 shots with energy of 100mJ and frequency of 15Hz with 15mm plastic tip, and for the tip slip, Neutral Thork® Lotion, RMC was used. Seven ESWT sessions were held, the average time of each was seven minutes, twice a week and the seventh session was held minutes before the surgical procedure of bariatric surgery, therapy was performed in an area of 150cm² on the left side of the abdominal region following the midline. The right side of the participants' abdomen did not receive ESWT and was termed as control.
  Arms: Treatment groupThorck Shock Wave Ibramed (terapia ESWT)- fat cell death

SUMMARY:
Informative Summary: Extracorporeal shockwave therapy (ESWT) is a new method for treating aesthetic disorders within the field of aesthetic medicine, its mechanisms of action and physiological effects promise to combat localized fat accumulation, improve skin appearance, favor neocolagenesis and neovascularization. There are currently few studies on ESWT that can claim this benefit, but therapy has been shown to be safe and does not generate adverse reactions to individuals.

Objective: To evaluate the physiological effects and mechanisms of ESWT acting on subcutaneous adipose tissue and adjacent structures through an experimental study.

Methods: A randomized experimental clinical study will be performed in 30 women with grade I, II and III obesity who participated in the multidisciplinary preoperative preparation group for bariatric surgery with previously scheduled surgery. Participants will receive ESWT application within hours of surgery, or in the weeks prior to bariatric surgery, during the surgical procedure a small sample of subcutaneous adipose tissue will be taken for histological and immunohistochemical analysis.

Hypotheses: Through histological and immunohistochemical analysis of the subcutaneous adipose tissue sample, the investigators can identify which real physiological effect and mechanism of action the ESWT has on subcutaneous adipose tissue, epidermis and adjacent structures, thus confirming the benefits of therapy.

Statistical analysis: A descriptive analysis of the results obtained in the histological analysis will be performed initially, with frequency tables for categorical and descriptive variables (mean, standard deviation, median, minimum and maximum values) for continuous or numerical variables. In order to compare the main variables between groups and session number, the analysis of variance (ANOVA) will be used for repeated measures. For comparison between groups the Tukey test will be used. The significance level adopted for the statistical tests will be 5% or p <0.05.

DETAILED DESCRIPTION:
ESWT procedures The participants received seven ESWT therapy sessions twice a week, the last session being about twenty minutes before the surgical procedure of bariatric surgery, the therapy was performed in an area of 150 cm² on the left side of the abdominal region, following the white line, frequently 15Hz, with 4,000,000 shots with 180mJ energy and 15mm stainless steel tip and 2,000,000 shots with 100mJ energy with 15mm plastic tip, for the tip slip a Thork ® Essential Cosmetics Industry Lotion was used LTDA- MED Anvisa nº 25351.419510 / 2017- 95.

For therapy, the THORK Shock Wave® equipment - IBRAMED- Industria Brasileira de Equipamentos Electromédicos EIRELI, approved by Anvisa nº 10360310036, was used.

The direct side of the participants' abdomen was used as a control and did not receive ESWT therapy.

Surgical procedure

After performing the anesthetic procedure at the beginning of the surgical act of bariatric surgery, the surgeon responsible removed two fragments of cutaneous tissue with an average size of 4 cm in diameter, one sample from the region previously demarcated on the left side of the abdomen and the other sample on the side contralateral where there was no demarcation considered as control.

Histological procedure After collection, the material was stored in a container with 10% formaldehyde for 48 hours. The samples were processed histotechnically, embedded in paraffin and then cut with a rotating microtome in sections of 3-5 μm thick.

For morphological evaluation of the cutaneous tissue and collagen cells, the slides were stained with Hematoxylin and Eosin (HE) and Masson's Trichrome (ab150686, Abcam, Cambridge, United Kingdom). The slides were evaluated by light microscopy with a binocular microscope (Nikon YS 100, Japan) adapted with a WSCF 10X / 18 eyepiece and Nikon 4X / 0.10, 10X / 0.25, 40X / 0.65 and 100X / 1 lenses, 25.

To differentiate the types of collagen fibers, Picrosirius Red staining (ab150681, Abcam) was used. After staining, the slides were analyzed under polarized light with a DMR microscope (Leica) and photographs were taken at 400 × magnification, the collagen fibers were differentiated by means of their staining and the type I collagen fibers were yellow-orange in color. some cases even red and type III with green coloring, to quantify the analyzes, the ImageJ® software (NIH, Bethesda, USA) was used.

All preparations were made following the protocol of antibodies and standardized by the laboratory of pathological analysis at Hospital de Clinicas da Unicamp.

Immunohistochemical procedures To perform immunohistochemical reactions, the paraffin blocks with the skin samples were cut to a thickness of 3 μm and placed on signed slides (3-aminopropyl-triethoxysilane, Sigma-Aldrich, USA). Positive and negative controls were performed in all reactions. The reactions were carried out according to previously published protocols

Briefly, the tissues were subjected to dewaxing, rehydration and endogenous peroxidase blocking processes. Antigenic recovery was performed with a solution of ethylenediamine tetraacetic acid (EDTA), pH 9.0, in an electric pressure cooker for 15 minutes.

For immunohistochemical analysis, the following antibodies, markers of fibroblast growth factors (FGFs) and their respective receptors were used: FGF1 (Antibody sc-55520, Santa Cruz Biotechnology, USA), FGF2 (Antibody sc-365106, Santa Cruz Biotechnology), FGFR1 (Antibody sc-121, Santa Cruz Biotechnology), FGFR2 (Antibody sc-122, Santa Cruz Biotechnology) and to evaluate cell proliferation, the marker Ki67 (Antibody ab92742, Abcam) was used.

The antigen-antibody reaction was developed using the chromogenic substrate (3.3 diaminobenzidine-DAB, Sigma-Aldrich). Then the slides were scanned and digitally analyzed also according to previous protocols

ELIGIBILITY:
Inclusion Criteria:

-

The study will include patients:

* female gender, over 18 years of age;
* With obesity grade I, II and III;
* Patient with surgical indication for bariatric surgery;
* Roux-en-Y gastric bypass type surgical procedure;
* Agree to participate and sign the consent form;

Exclusion Criteria:

* Male gender;
* smoking;
* cognitive limitations
* Carriers diabetes mellitus;
* Performed aesthetic treatment on the abdomen in the last month;
* Patients with skin lesions such as dermatitis and dermatosis;
* Patients with acute deep vein thrombosis (DVT);
* About or near cancerous lesions;
* Patients with cardiac pacemakers or other implanted electronic devices.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with obesity
Enrollment: 10 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical procedures | one month
  Immunohistochemical reactions were performed on 3μm-thick sections, arranged on silanized slides. The antibodies used were: polyclonal anti-Caspase3 , monoclonal anti-Cleaved Caspase 3 ; monoclonal anti-CD68, monoclonal anti-hormone-sensitive lipase - HSL - and Adipophilin. After preparing the slides, they were analyzed with a DMR microscope (Leica), and photographs were taken at 400x magnification. To quantify the analyses, the ImageJ® software (NIH, Bethesda, USA) was used.
  All reactions were performed following the manufacturers' protocol and all were standardized by the pathological analysis laboratory of the Hospital de Clínicas da Unicamp. The quantification of immunostaining was performed considering the number of positive cells and intensity, with final scores ranging from 0-300

CONTACTS AND LOCATIONS:
Overall Officials: Debora Modena, Dr, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Unicamp, Campinas, São Paulo, Brazil